CLINICAL TRIAL: NCT00656110
Title: Randomized, Placebo-Controlled Trial of Bilateral 3rd/4th Common Digital Foot Nerve Injections to Treat Restless Legs Syndrome
Brief Title: Neuroma Injections to Treat Restless Legs Syndrome - RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lowcountry Infectious Diseases (Other)
Responsible Party: Ludwig A. Lettau, M.D., Lowcountry Infectious Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LID-RLS-RCT-01
Record Dates: First submitted 2008-04-06; First posted 2008-04-10 (Estimated); Last update posted 2009-03-10 (Estimated); Status verified 2009-03

CONDITIONS: Restless Legs Syndrome
Keywords: Restless legs syndrome; Morton's neuroma; Randomized controlled trial
MeSH Terms: conditions — Restless Legs Syndrome; Morton Neuroma | interventions — Ethanol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-T (Experimental): Treatment Group
  Interventions: Drug: equal parts of 0.5% plain Marcaine and 2% lidocaine mixed with 0.8 mg Depo-medrol/4% absolute alcohol in a total injection volume of 1 ml
- 2-P (Placebo Comparator): Placebo comparator
  Interventions: Drug: Normal saline - 1ml

INTERVENTIONS:
Drug: equal parts of 0.5% plain Marcaine and 2% lidocaine mixed with 0.8 mg Depo-medrol/4% absolute alcohol in a total injection volume of 1 ml — Bilateral 3rd/4th common digital nerve injections with neuroma treatment mixture given weekly for 3 weeks
  Arms: 1-T
Drug: Normal saline - 1ml — Bilateral 3rd/4th common digital nerve injections with normal saline given weekly for 3 weeks
  Arms: 2-P

SUMMARY:
The purpose of this study is to determine whether, in a randomized, placebo-controlled trial, restless legs syndrome (RLS) can be caused by pinched and damaged foot nerves called neuromas.

DETAILED DESCRIPTION:
Restless legs syndrome (RLS) is a medical condition in which there is an almost irresistible urge to move the legs in response to uncomfortable, difficult-to-describe leg sensations that are usually worse in the evening and especially noticeable when inactive such as sitting in a chair watching TV or when resting in bed trying to go to sleep or back to sleep after awakening. Most patients with RLS, while asleep, also have involuntary leg movements called periodic limb movements of sleep (PLMS). During a sleep study, brain wave monitoring of patients with RLS/PLMS often shows that the nighttime leg movements are associated with brain stimulation and arousal to a lighter stage of sleep. When many such brain arousals happen through the night, the natural pattern of deep sleep may be severely disrupted. Such disturbed sleep is of poorer quality and is less refreshing. The combination of RLS-related delay of initiation or resumption of sleep and PLMS-related poor quality of sleep may result in a severe sleep disorder manifested by morning sluggishness and increased daytime fatigue. The cause(s) of RLS and PLMS have not been determined. Neurologists believe that they originate in the brain in areas that control movement and may be related to localized low levels of dopamine (a chemical messenger between nerve cells) or related to disordered brain iron metabolism, but these theories have never been proven.

RLS and PLMS generally are lifelong conditions for which there is no cure. RLS is treated with medications targeting the brain and categories of drugs that have been used to treat symptoms (with varying success) include mainly dopaminergic drugs but also sedatives, anti-seizure drugs, and pain medications such as narcotics. Two dopaminergic drugs have been approved by the FDA for the treatment of RLS: ropinirole ("Requip") in 2005 and pramipexole ("Mirapex") in 2006. However such drugs are far from ideal because, in addition to the problem of side effects, some patients may not respond to these drugs or symptoms may only partially improve. Also, any improvement only occurs while continuing to take the drug, and finally, symptoms may sometimes become much worse after an initial period of improvement, a phenomenon called augmentation.

Foot neuromas are nerve entrapments ("pinched nerves") which form at points where the common interdigital nerves must stretch under ligaments between the metatarsal heads in the ball of each foot. Repeated irritation and damage to the nerves at those stretch points eventually results in fibrous thickening and enlargement of the nerve tissue into a lump called a neuroma. This most commonly involves a nerve in the ball of the foot between the third and fourth toes ("Morton's Neuroma"), but neuromas also often form at the entrapment/stretch point of the nerves between the second/third and fourth/fifth toes.

Neuromas may be completely asymptomatic in the foot or may cause variable degrees of unilateral or bilateral foot pain and numbness brought on or made worse by tight shoes, high heels, or prolonged walking or standing. When neuromas become more severely symptomatic, they may cause neuropathic symptoms such as burning, tingling, numbness, electric shock shooting pains, and hypersensitivity. Neuromas are treated with a series of injections (local anesthetic combined with either steroids and/or alcohol solution) given into the neuroma-containing space in the ball of the foot. It is believed that these injections serve to calm the nerve irritability which usually results in improvement or sometimes even complete resolution of the neuropathic symptoms (burning pain, etc.).

Previous studies by our group determined that many patients with neuropathic foot symptoms (burning, tingling, electric shocks, numbness, etc.) who had been previously diagnosed with "peripheral neuropathy," actually had neuromas in both feet as the cause of their symptoms. The causative role of neuromas in these patients was demonstrated by the fact that their chronic pain symptoms improved (in some cases markedly so) with standard neuroma injection treatment. In addition to improvement in their neuropathic foot pains, many patients also reported that they were sleeping much better. Such patients reported not only a decrease in their RLS-type leg restlessness but also that their spouse had noted a decrease in their PLMS-type nighttime leg movements, all as a direct result of their bilateral neuroma injections. These reports prompted further study of patients who had RLS/PLMS both with and without neuropathic foot pains.

Most patients with RLS/PLMS do not have major foot complaints. However such patients have been consistently found by us to have physical evidence of neuromas on examination of their feet and standard treatment of their bilateral neuromas usually resulted in prompt improvement of the symptoms related to RLS/PLMS along with the quality of their sleep. 15 such patients were studied intensively before and after neuroma treatment and 9 of these patients had complete relief of RLS symptoms for an average of over 2 months after a series of neuroma injections (Lettau LA, Gudas CJ. Bilateral Morton's neuromas as an etiology of restless legs syndrome. J SC Med Assoc 2005; 101: e341-e347).

However, the prevailing theory remains that RLS is of brain origin, so that a controlled study is being done to further support a foot neuroma origin of RLS by comparing the responses of two randomized groups of adults with RLS - one group to receive a series of 3 bilateral neuroma treatments (equal parts of 0.5% plain Marcaine and 2% lidocaine mixed with 0.8 mg Depo-medrol/4% absolute alcohol in a total injection volume of 1 ml injected weekly over 3 weeks) and a second "control" group to receive only placebo (normal saline) injections over a similar time period. Neither group will be told whether they are getting the actual treatment solution or placebo over the 3 weeks. After the 3 weeks are up, the patients who had received the placebo, will be told of their status and will be given the real injection treatments over the next 3 weeks. One follow-up visit (4 weeks after the last treatment injection) is planned to assess short term duration of treatment(s).

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms (that fulfill the 4 essential clinical criteria for RLS) of at least 6 months duration with a current IRLS-rs score indicative of at least moderate severity (15 or greater)
* Evidence of bilateral 3rd/4th interspace neuromas by both physical examination and ultrasound criteria at initial evaluation
* Willingness and ability of patient to participate in initial weekly evaluation/neuroma treatment visits and subsequent periodic follow-up visits over a period of approximately 6-9 weeks.
* Off dopaminergic drug treatment (ropinirole-"Requip" or pramipexole-"Mirapex") starting 2 weeks prior to the initial foot injections and for the duration of the study.

Exclusion Criteria:

* Major foot deformity, previous major foot surgery, or previous neuroma injections
* Known or suspected obstructive sleep apnea
* Allergy to any of injection components (depo-medrol, lidocaine, marcaine, absolute alcohol)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-11 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
International Restless Legs Rating Scale | Weekly during the study and three weeks after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig A Lettau, MD, Principal Investigator — Lowcountry Infectious Diseases
Locations (1):
- Southeastern Foot Specialists, Charleston, South Carolina, United States

REFERENCES:
- [Background] Lettau LA, Gudas CJ. Bilateral Morton's neuromas as an etiology of restless legs syndrome. Journal of the South Carolina Medical Association 101: e341-e347, 2005